CLINICAL TRIAL: NCT01709292
Title: Pharmacodynamic Study of Vemurafenib in the Neoadjuvant Setting in Patients With Locally Advanced Thyroid Cancer
Brief Title: Vemurafenib Neoadjuvant Trial in Locally Advanced Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0471; NCI-2012-02171 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-07-25; First posted 2012-10-18 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; ERK; Extracellular-signal-regulated kinase; Biomarkers; Papillary thyroid cancer; PTC; BRAF mutated; Vemurafenib; PLX4032; RO5185426; Zelboraf™
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary | interventions — Vemurafenib; Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vemurafenib - (Presurgery) (Experimental): All Groups: Vemurafenib 960 mg by mouth 2 times a day for 56 days prior to surgery (patients not planned for surgical resection will have a core biopsy at day 56 +/- 7 days).
  Interventions: Drug: Vemurafenib (All Groups); Drug: Vemurafenib (Post Surgery) - Group A + C; Other: Post Surgery - Group B
- Vemurafenib (Post Surgery) - Group A (Experimental): Vemurafenib 960 mg by mouth two times a day 2 weeks post-surgery, or if patients have not sufficiently recovered at that point, as soon as their condition permits. Patients in Group A restaged 8 weeks after resuming drug. If patients in Group A demonstrate either stable or regressing disease, they will continue on vemurafenib with restaging occurring every 8 weeks until no longer benefitting from the drug.
  Interventions: Drug: Vemurafenib (Post Surgery) - Group A + C
- Post Surgery - Group B (No Intervention): Post Surgery - Group B: Patients discontinue vemurafenib after surgery but will be restaged with CT neck 8 weeks after surgery.
- Vemurafenib - Group C (Experimental): Patients not scheduled for surgical resection undergo a CT scan and core biopsy at day 56, Vemurafenib 960 mg by mouth twice a day unless there is evidence of progressive disease on day 56 CT scan. Patients evaluated for resectability after each CT scan is performed. If scheduled for resection, patient continues vemurafenib until surgery and follows same treatment schema as patients in Groups A and B.
  Interventions: Drug: Vemurafenib (Post Surgery) - Group A + C

INTERVENTIONS:
Drug: Vemurafenib (All Groups) — 960 mg by mouth 2 times a day 56 days prior to surgery (patients not planned for surgical resection will have a core biopsy at day 56.
  Other Names: PLX4032; RO5185426; Zelboraf™
  Arms: Vemurafenib - (Presurgery)
Drug: Vemurafenib (Post Surgery) - Group A + C — Group A: 960 mg by mouth twice a day 2 weeks post-surgery. Restaged 8 weeks after resuming drug. If patients demonstrate either stable or regressing disease, they will continue on vemurafenib with restaging occurring every 8 weeks until they are no longer benefitting from the drug.
  Group C: Patients not scheduled for surgical resection undergo a CT scan and core biopsy at day 56. Vemurafenib 960 mg by mouth twice a day, continued unless there is evidence of progressive disease on day 56 CT scan. Patients restaged every 8 weeks and continue vemurafenib until no longer benefitting from the drug. Patients evaluated for resectability after each CT scan is performed. If patient is scheduled for resection, then patient will continue vemurafenib until surgery and will follow the same treatment schema as patients in Groups A and B.
  Other Names: PLX4032; RO5185426; Zelboraf™
  Arms: Vemurafenib (Post Surgery) - Group A; Vemurafenib - (Presurgery); Vemurafenib - Group C
Other: Post Surgery - Group B — Patients who have had a complete surgical resection, and who do not have evidence of metastatic disease will discontinue vemurafenib after surgery. Patients restaged with CT neck 8 weeks after surgery.
  Arms: Vemurafenib - (Presurgery)

SUMMARY:
The goal of this clinical research study is to learn about how vemurafenib may affect certain biomarkers in patients with PTC. Biomarkers are in the blood/tissue and may be related to your reaction to the study drug. The safety of this drug will also be studied.

Vemurafenib is designed to block the BRAF gene mutation. This mutation causes cancer and cancer growth. By blocking this mutation, the drug may kill the cancer cells with the mutation and/or stop the tumor from growing.

DETAILED DESCRIPTION:
Study Drug Administration and Groups:

If you are found to be eligible to take part in this study, you will take 4 tablets of vemurafenib by mouth 2 times each day for 56 days. You should take each dose about 12 hours apart. If you miss taking the drug at a scheduled time by more than 4 hours, you should skip that dose and wait until the next dose.

After 56 days, the treatment you receive will depend on what group you are assigned to:

* If the disease has spread outside the neck, you will be in Group A.
* If the disease is able to be entirely removed through surgery, you will be in Group B.
* If the disease is unable to be operated on, you will be in Group C.

Study Visits:

At all visits, you will be asked about any side effects you may be having and about any other drugs you may be taking.

Before you take the study drug (Baseline):

* You will have a procedure called a laryngoscopy, in which a tube with a small camera in inserted into the nose to inspect your sinus, throat, and voice box.
* You will have a colonoscopy if you have a history of abnormal growth in the bowel (polyps or colon cancer). During this procedure a tube with a small camera is inserted in the anus to inspect your large bowel.

At Day 28:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will have an EKG.
* Blood (about 1 tablespoon) will be drawn for routine tests.

Within 1 week before Day 56, you will have CT scans of the neck, chest, and abdomen to check the status of the disease.

At Day 56, if you are in Group A or B, you will have surgery to remove the tumor. You will sign a separate consent form that describes this surgery and its risks. If you are in Group C, you will have a core biopsy. During the surgery/biopsy, blood (about 1 teaspoon) will also be collected for biomarker testing.

Follow-Up:

Your follow-up after the surgery/biopsy will depend on which study group you are in.

Groups A and C:

If you are in Group A, you will stop taking the study drug for about 2-4 weeks after you have surgery. If you are in Group C, you will not stop taking the study drug. Every 4 weeks (after you resume taking the study drug if you are in Group A, and after the biopsy if you are in Group C):

* You will have a physical exam, including measurement of your vital signs and a skin exam.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any other drugs you may be taking and about any side effects you may be having.
* If you are in Group A, these tests will also be performed the day you start taking the study drug again. You will also have an EKG.

Additionally, every 8 weeks (if you are in Group A or C), you will have CT scans of the neck, chest, and abdomen to check the status of the disease. Blood (about 1 teaspoon) will also be drawn for biomarker testing at the first of these visits.

About 1 year after your laryngoscopy and colonoscopy, these procedures will be performed again to check for side effects related to the study drug. If you did not receive a baseline colonoscopy, this procedure will be performed about 1 year after starting vemurafenib. If you continue on study drug for more than a year, you will have a laryngoscopy every 12 months.

At any time the study doctor thinks it is needed, you will have a colonoscopy and laryngoscopy.

About 1 year after the surgery/biopsy, you will return to clinic to check if the disease has come back. At this visit, you will have a CT scan or ultrasound of the neck, and blood (about 1 tablespoon) will be drawn for tests of your thyroid function.

If after 4 months the study doctor thinks it is in your best interest, you will only need to have study visits every 8 weeks. You will still have blood (about 1 tablespoon) drawn for routine tests at a local lab and you will be called by the study staff to check on you. Each call will last about 5-10 minutes.

If you are in Group C, and if during follow-up the study doctor decides that the disease can be operated on, you will be crossed over to Group A or B. You will have surgery and have the follow-up visits described for that study group.

Group B:

If you are in Group B, you will have a follow-up visit about 2 weeks after surgery. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any other drugs you may be taking and about any side effects you may be having.

You will have a second follow-up visit about 8 weeks after surgery. You will have a CT scan of the neck to check the status of the disease. You will have the option of continuing to receive vemurafenib if your doctor thinks it is in your best interest. If you do continue on vemurafenib, you will follow the Group A follow-up schedule (above).

About 1 year after your laryngoscopy and colonoscopy, these procedures will be performed again to check for side effects related to the study drug. If you did not receive a baseline colonoscopy, this procedure will be performed about 1 year after starting vemurafenib.

At any time the study doctor thinks it is needed, you will have a colonoscopy and laryngoscopy.

About 1 year after the surgery/biopsy, you will return to clinic to check if the disease has come back. At this visit, you will have a CT scan or ultrasound of the neck, and blood (about 1 tablespoon) will be drawn for tests of your thyroid function.

Length of Study:

If you are in Group A or C, you will continue to take the study drug for as long as the study doctor thinks it is in your best interest. If you are in Group B, you will take the study drug for 56 days and will no longer take it after surgery. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over when you have completed the follow-up visits.

End-of-Study Visit/Call:

After you stop taking the study drug, you will have an end-of-study visit or phone call. You will be asked about any other drugs you may be taking and about any side effects you may have had. If you are called, the call will last about 5-10 minutes.

This is an investigational study. Vemurafenib is FDA approved and commercially available for the treatment of late-stage melanoma. It is investigational to use this drug to treat thyroid cancer.

Up to 22 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Primary papillary thyroid cancer (PTC), which appears to be stage T3 or T4 on imaging or with macroscopic lymph node involvement AND requires surgical resection.
2. Persistent or locally recurrent PTC with macroscopic lymph node involvement which requires surgical resection.
3. Patients deemed inoperable (no scheduled surgery) are eligible for this trial, as they could be surgical candidates after treatment with vemurafenib. Inoperable patients must be naïve to therapies targeting the MAPK pathway.
4. BRAF V600E mutation detected in the primary tumor or the recurrent/persistent tumor.
5. Total bilirubin </= 1.5 x upper limit of normal (ULN). Patients with Gilbert's syndrome are excluded from this requirement. Aspartate transaminase (serum glutamic oxaloacetic transaminase) / alanine transaminase (serum glutamic pyruvic transaminase) (AST[SGOT]/ALT[SGPT]) </= 2.5 x ULN, (5 x ULN for patients with concurrent liver metastases). Serum creatinine </= within 1.5 x ULN. Absolute neutrophil count (ANC) >/= 1.0 x 10^9/L; platelets >/= 100 x 10^9/L, HgB>9 mg/dL
6. Antiangiogenic therapy, specifically vascular endothelial growth factor (VEGF) and VEGF receptor (VEGFR) inhibitors, can interfere with wound healing and therefore will only be allowed if the agent has been discontinued for at least 14 days prior to day 1. Group C patients must be naïve to therapies which target mitogen-activated protein kinase (MAPK).
7. Ability to swallow pills.
8. Eastern Cooperative Oncology Group (ECOG) performance status </= 2
9. Age >/= 18
10. Ability to provide consent.

Exclusion Criteria:

1. Histological diagnosis other than PTC. Patients with anaplastic tumors are not eligible. However, patients whose tumors contain areas of un-differentiated or dedifferentiated histology may enroll provided the original diagnosis was clearly PTC, and the tumor histology remains predominantly papillary at enrollment.
2. Refractory nausea and vomiting, malabsorption, or significant bowel resection that would preclude adequate absorption.
3. Known hepatitis B or C virus (HBV or HCV) infection, unless the patient has been cleared for chemotherapy from experts on viral hepatitis (infectious disease specialists or hepatologists).
4. Pregnant or lactating women. All pre-menopausal women being screened must have a negative serum pregnancy test within 14 days prior to commencement of dosing. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for >/= 1 year
5. Untreated brain metastases.
6. Chemotherapy or targeted therapy within 14 days or 5 half-lives (whichever is longer) prior to the start of study treatment.
7. Patients with history of long QT syndrome, uncorrectable electrolyte abnormalities, or QTc>500msec.
8. History of significant cardiac disease or uncontrolled arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in ERK (Extracellular-Signal-Regulated Kinase) Phosphorylation and Tumor Size | 56 days
  ERK phosphorylation and tumor size measured at baseline before first dose of Vemurafenib and again after 56 days of Vemurafenib. We will test whether correlation between percent change in ERK phosphorylation and percent change in tumor size is different from 0 with a t-test.

SECONDARY OUTCOMES:
Objective Response Rate | 56 days
  Objective response rate defined as proportion of patients who have had a partial response (PR) or complete response (CR) after initiation of therapy with Vemurafenib, using RECIST 1.1. All patients who complete baseline and day 56 scans evaluable for this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E. Cabanillas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org